CLINICAL TRIAL: NCT02524652
Title: Postoperative Analgesic Efficacy of Local Infiltration Analgesia Versus Adductor Canal Block After Anterior Cruciate Ligament Reconstruction: A Randomised Controlled Double-blinded Trial
Brief Title: Local Infiltration Analgesia vs Adductor Canal Block for Analgesia After Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, Program Director, Regional Anaesthesia, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CER 193-15
Record Dates: First submitted 2015-08-06; First posted 2015-08-17 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Rupture of Anterior Cruciate Ligament; Infiltration; Regional Anesthesia Morbidity
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local infiltration analgesia (Experimental): Infiltration of the knee by the surgeon with local anaesthetics under general anaesthesia.
  Interventions: Drug: Ropivacaine 0.5% 20 mLs
- Adductor canal block (Active Comparator): Injection of local anaesthetics under ultrasound guidance in the adductor canal by the anaesthesiologist after the surgery, before awaking the patient.
  Interventions: Drug: Ropivacaine 0.5% 20 mLs

INTERVENTIONS:
Drug: Ropivacaine 0.5% 20 mLs — Injection of the local anesthetic at the end of surgery, either in the surgical sites by the surgeon, or in the adductor canal block by the anesthesiologist under ultrasound guidance.
  Other Names: Naropine, Naropin

SUMMARY:
Early rehabilitation after anterior cruciate ligament reconstruction is of paramount importance and requires optimal pain control based on a multimodal concept, including injection of local anaesthetics. Regarding this latter, different options have emerged recently such as the adductor canal block, performed before the surgery by the anaesthesiologist or the infiltration of the articulation performed by the surgeon at the of the intervention. No trial has compared these two approaches. As practice of medicine should be based on evidence, we decided to undertake this randomised controlled trial where we compared the adductor canal block with the local infiltration analgesia technique in terms of pain and functional outcomes

DETAILED DESCRIPTION:
Patients scheduled to undergo anterior cruciate ligament reconstruction under general anaesthesia will be randomly allocated to two groups: local infiltration analgesia or adductor canal block.

The local infiltration analgesia will be performed by the surgeon at the end of surgery with 20 mLs of ropivacaine 0.5%. The adductor canal block will be performed by the anaesthesiologist under ultrasound guidance after the surgery, before awaking the patient, using the same solution (20 mLs ropivacaine 0.5%)

Postoperative analgesia will include intravenous patient-controlled analgesia of morphine (settings 1 mg/ml, 2 ml/10 minutes, 40 mg/4 hours), ibuprofen (3x400 mg) and acetaminophen (4x1000 mg).

A research assistant and a physiotherapist, both blinded to the group allocation, will collect pain and rehabilitation data, respectively.

ELIGIBILITY:
Inclusion Criteria:

* patients from 18 to 50 years old scheduled to undergo anterior cruciate ligament reconstruction

Exclusion Criteria:

* peripheral neuropathy
* pre-existing femoral neuropathy
* diabetes mellitus
* alcoholism
* drug addiction
* cancer with chemotherapy
* chronic pain state

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2015-09; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption (mg) | 24 h postoperatively

SECONDARY OUTCOMES:
Total morphine consumption (mg) | 2 h postoperatively
Total morphine consumption (mg) | 48 h postoperatively
Total morphine consumption (mg) | 72 h postoperatively
Pain scores (numeric rating scale, 0-10) at rest and on movement | 2 h postoperatively
Pain scores (numeric rating scale, 0-10) at rest and on movement | 12 h postoperatively
Pain scores (numeric rating scale, 0-10) at rest and on movement | 24 h postoperatively
Pain scores (numeric rating scale, 0-10) at rest and on movement | 36 h postoperatively
Pain scores (numeric rating scale, 0-10) at rest and on movement | 48 h postoperatively
Pain scores (numeric rating scale, 0-10) at rest and on movement | 60 h postoperatively
Pain scores (numeric rating scale, 0-10) at rest and on movement | 72 h postoperatively
Postoperative nausea and vomiting (yes/no) | 24 h postoperatively
Postoperative nausea and vomiting (yes/no) | 48 h postoperatively
Postoperative nausea and vomiting (yes/no) | 72 h postoperatively
Pruritus (yes/no) | 24 h postoperatively
Pruritus (yes/no) | 48 h postoperatively
Pruritus (yes/no) | 72 h postoperatively
Active flexion | 24 h postoperatively
  Flexion of the knee by the patient measured in degrees
Active flexion | 48 h postoperatively
  Flexion of the knee by the patient measured in degrees
Active flexion | 72 h postoperatively
  Flexion of the knee by the patient measured in degrees
Quadriceps muscle strength (numeric scale, 1-5) | 24 h postoperatively
Quadriceps muscle strength (numeric scale, 1-5) | 48 h postoperatively
Quadriceps muscle strength (numeric scale, 1-5) | 72 h postoperatively
Distance walked (meters) | 24 h postoperatively
Distance walked (meters) | 48 h postoperatively
Distance walked (meters) | 72 h postoperatively
Anterior Cruciate Ligament - Return to Sport after Injury scale | 4 months postoperatively
Anterior cruciate ligament -Return to Sport after Injury scale | 8 months postoperatively
International Knee Documentation Committee score | 4 months postoperatively
International Knee Documentation Committee score | 8 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Eric Albrecht, PD Dr, Principal Investigator — CHUV
Locations (1):
- Department of Anesthesia, Centre Hospitalier Universitaire Vaudois and University of Lausanne, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Stebler K, Martin R, Kirkham KR, Lambert J, De Sede A, Albrecht E. Adductor canal block versus local infiltration analgesia for postoperative pain after anterior cruciate ligament reconstruction: a single centre randomised controlled triple-blinded trial. Br J Anaesth. 2019 Aug;123(2):e343-e349. doi: 10.1016/j.bja.2019.04.053. Epub 2019 May 24. PMID 31130273